CLINICAL TRIAL: NCT05154175
Title: Effectiveness of Ottobock Helmet Therapy in Infants With Plagiocephaly, Brachycephaly or Combination of Both and Parents' Satisfaction
Brief Title: Effectiveness of Ottobock Helmet Therapy in Infants With Plagiocephaly, Brachycephaly or Combination of Both
Status: Completed | Type: Observational
Sponsor: Otto Bock France SNC (Industry)
Collaborators: Quanta Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: BP-11-PT006-FR-01-2108
Record Dates: First submitted 2021-11-15; First posted 2021-12-10 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Plagiocephaly, Positional; Plagiocephaly, Nonsynostotic; Brachycephaly
Keywords: Cranial orthosis; Helmet treatment
MeSH Terms: conditions — Plagiocephaly, Nonsynostotic; Craniosynostoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Ottobock helmet: Infants treated with an Ottobock helmet
  Interventions: Device: Ottobock helmet

INTERVENTIONS:
Device: Ottobock helmet — Patients treated in current practice
  Other Names: MyCRO Band

SUMMARY:
The objective of the research is to measure the effectiveness of the Ottobock helmet, an innovative 3D-printed cranial orthosis used to correct infant cranial positional deformation: plagiocephaly, brachycephaly or combination of both.

This research is a retrospective multi-centric study composed of a collection of clinical data from orthotists database and a survey for patient's parents.

DETAILED DESCRIPTION:
The Ottobock helmet is a cranial orthosis used to correct infant cranial positional deformation: plagiocephaly, brachycephaly or combination of both. This medical device is a 3D-printed helmet, with an elastic closing system which allow the head growth, maintain a constant pressure in the helmet and ensure a good adjustment.

Even though there is an effectiveness observed, there are no existing clinical evidences on this type of helmet so far, and there is a need to conduct a research on a large number of patients to measure the effectiveness and describe the population treated. This study will give more information to health professionals (doctors, orthopedic technicians, etc.) and health authorities, about the benefits of the orthopedic treatment of the positional cranial deformations in infants.

The study is composed of an electronic case report form (eCRF) to be fulfilled by the orthotists and an electronic questionnaire (ePRO) to be fulfilled by the patient's parents. The electronic questionnaires, data treatment and analysis are handled by a Contract Research Organization (CRO).

ELIGIBILITY:
Inclusion Criteria:

* Infant with positional cranial deformation
* Infant treated with an Ottobock helmet between May 1st, 2020 and May 1st, 2021

Exclusion Criteria:

* Patient whose parents (or legal guardians) disagree to participate in the study.
* Patient whose parents (or legal guardians) are unable to understand or answer the questionnaire.

Ages: 3 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population is composed of infants who have been fitted with an Ottobock helmet to treat their positional cranial deformation: plagiocephaly, brachycephaly or a combination of these two deformations.
Sampling Method: Probability Sample
Enrollment: 452 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Cranial deformation index | 6 weeks
  The cranial deformation index is a ratio (%) of head diameters characterizing head deformation.

SECONDARY OUTCOMES:
Satisfaction of parents regarding the device and the services provided by the orthotist | Through study completion, an average of 6 months
  QUEST 2.0

CONTACTS AND LOCATIONS:
Overall Officials: Hannelore Willenborg, Dr., Study Chair — Hannover University Hospital Center, Diakovere Annastift, Germany; Dorothea Daentzer, Prof.Dr.med., Study Chair — Hannover University Hospital Center, Diakovere Annastift, Germany
Locations (12):
- France (12):
  - Chabloz Orthopédie Annecy, Annecy
  - Orthèse Prothèse Changeant OPC, Castelnau-le-Lez
  - Chabloz Orthopédie Clermont-Ferrand, Cournon-d'Auvergne
  - Technic'Ortho, Lay-Saint-Christophe
  - Chabloz Orthopédie Nice, Nice
  - Chabloz Orthopédie Lyon, Oullins
  - Orthèses Prothèses Générales OPG, Paris
  - Chabloz Orthopédie Valence, Portes-lès-Valence
  - Chabloz Orthopédie Dijon, Saint-Apollinaire
  - Chabloz Orthopédie Grenoble, Seyssinet-Pariset
  - Chabloz Orthopédie Toulouse, Toulouse
  - Chabloz Orthopédie Venelles, Venelles

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Argenta L, David L, Thompson J. Clinical classification of positional plagiocephaly. J Craniofac Surg. 2004 May;15(3):368-72. doi: 10.1097/00001665-200405000-00004. PMID 15111792
- [Background] van Vlimmeren LA, Takken T, van Adrichem LN, van der Graaf Y, Helders PJ, Engelbert RH. Plagiocephalometry: a non-invasive method to quantify asymmetry of the skull; a reliability study. Eur J Pediatr. 2006 Mar;165(3):149-57. doi: 10.1007/s00431-005-0011-1. Epub 2005 Oct 7. PMID 16211401
- [Background] Graham JM Jr, Gomez M, Halberg A, Earl DL, Kreutzman JT, Cui J, Guo X. Management of deformational plagiocephaly: repositioning versus orthotic therapy. J Pediatr. 2005 Feb;146(2):258-62. doi: 10.1016/j.jpeds.2004.10.016. PMID 15689920
- [Background] Moss SD. Nonsurgical, nonorthotic treatment of occipital plagiocephaly: what is the natural history of the misshapen neonatal head? J Neurosurg. 1997 Nov;87(5):667-70. doi: 10.3171/jns.1997.87.5.0667. PMID 9347972
- [Background] Wendling-Keim DS, Mace Y, Lochbihler H, Dietz HG, Lehner M. A new parameter for the management of positional plagiocephaly: the size of the anterior fontanelle matters. Childs Nerv Syst. 2020 Feb;36(2):363-371. doi: 10.1007/s00381-019-04215-y. Epub 2019 Jun 17. PMID 31209640
- [Background] Loveday BP, de Chalain TB. Active counterpositioning or orthotic device to treat positional plagiocephaly? J Craniofac Surg. 2001 Jul;12(4):308-13. doi: 10.1097/00001665-200107000-00003. PMID 11482615
- [Background] Yoo HS, Rah DK, Kim YO. Outcome analysis of cranial molding therapy in nonsynostotic plagiocephaly. Arch Plast Surg. 2012 Jul;39(4):338-44. doi: 10.5999/aps.2012.39.4.338. Epub 2012 Jul 13. PMID 22872837
- [Background] Kim JK, Kwon DR, Park GY. A new ultrasound method for assessment of head shape change in infants with plagiocephaly. Ann Rehabil Med. 2014 Aug;38(4):541-7. doi: 10.5535/arm.2014.38.4.541. Epub 2014 Aug 28. PMID 25229033
- [Background] Holowka MA, Reisner A, Giavedoni B, Lombardo JR, Coulter C. Plagiocephaly Severity Scale to Aid in Clinical Treatment Recommendations. J Craniofac Surg. 2017 May;28(3):717-722. doi: 10.1097/SCS.0000000000003520. PMID 28468155
- [Background] Wilbrand JF, Schmidtberg K, Bierther U, Streckbein P, Pons-Kuehnemann J, Christophis P, Hahn A, Schaaf H, Howaldt HP. Clinical classification of infant nonsynostotic cranial deformity. J Pediatr. 2012 Dec;161(6):1120-5. doi: 10.1016/j.jpeds.2012.05.023. Epub 2012 Jun 23. PMID 22727872
- [Background] Graham JM Jr, Kreutzman J, Earl D, Halberg A, Samayoa C, Guo X. Deformational brachycephaly in supine-sleeping infants. J Pediatr. 2005 Feb;146(2):253-7. doi: 10.1016/j.jpeds.2004.10.017. PMID 15689919
- [Background] Kelly KM, Joganic EF, Beals SP, Riggs JA, McGuire MK, Littlefield TR. Helmet Treatment of Infants With Deformational Brachycephaly. Glob Pediatr Health. 2018 Oct 16;5:2333794X18805618. doi: 10.1177/2333794X18805618. eCollection 2018. PMID 30349871
- [Background] Hinken L, Willenborg H, Davila LA, Daentzer D. Outcome analysis of molding helmet therapy using a classification for differentiation between plagiocephaly, brachycephaly and combination of both. J Craniomaxillofac Surg. 2019 May;47(5):720-725. doi: 10.1016/j.jcms.2019.01.011. Epub 2019 Jan 17. PMID 30733135
- [Background] Schaaf H, Malik CY, Streckbein P, Pons-Kuehnemann J, Howaldt HP, Wilbrand JF. Three-dimensional photographic analysis of outcome after helmet treatment of a nonsynostotic cranial deformity. J Craniofac Surg. 2010 Nov;21(6):1677-82. doi: 10.1097/SCS.0b013e3181f3c630. PMID 21119399
- [Background] Hutchison BL, Hutchison LA, Thompson JM, Mitchell EA. Quantification of plagiocephaly and brachycephaly in infants using a digital photographic technique. Cleft Palate Craniofac J. 2005 Sep;42(5):539-47. doi: 10.1597/04-059r.1. PMID 16149837
- [Background] Wilbrand JF, Wilbrand M, Pons-Kuehnemann J, Blecher JC, Christophis P, Howaldt HP, Schaaf H. Value and reliability of anthropometric measurements of cranial deformity in early childhood. J Craniomaxillofac Surg. 2011 Jan;39(1):24-9. doi: 10.1016/j.jcms.2010.03.010. Epub 2010 Apr 24. PMID 20418107
- [Background] Purnell CA, Benz AW, Gosain AK. Assessment of Head Shape by Craniofacial Teams: Structuring Practice Parameters to Optimize Efficiency. J Craniofac Surg. 2015 Sep;26(6):1808-11. doi: 10.1097/SCS.0000000000001948. PMID 26267560
- [Background] Skolnick GB, Naidoo SD, Nguyen DC, Patel KB, Woo AS. Comparison of Direct and Digital Measures of Cranial Vault Asymmetry for Assessment of Plagiocephaly. J Craniofac Surg. 2015 Sep;26(6):1900-3. doi: 10.1097/SCS.0000000000002019. PMID 26267578
- [Background] Kluba S, Kraut W, Reinert S, Krimmel M. What is the optimal time to start helmet therapy in positional plagiocephaly? Plast Reconstr Surg. 2011 Aug;128(2):492-498. doi: 10.1097/PRS.0b013e31821b62d6. PMID 21788840
- [Background] Mulliken JB, Vander Woude DL, Hansen M, LaBrie RA, Scott RM. Analysis of posterior plagiocephaly: deformational versus synostotic. Plast Reconstr Surg. 1999 Feb;103(2):371-80. doi: 10.1097/00006534-199902000-00003. PMID 9950521
- [Background] Steinberg JP, Rawlani R, Humphries LS, Rawlani V, Vicari FA. Effectiveness of conservative therapy and helmet therapy for positional cranial deformation. Plast Reconstr Surg. 2015 Mar;135(3):833-842. doi: 10.1097/PRS.0000000000000955. PMID 25415272
- [Background] Kelly KM, Littlefield TR, Pomatto JK, Manwaring KH, Beals SP. Cranial growth unrestricted during treatment of deformational plagiocephaly. Pediatr Neurosurg. 1999 Apr;30(4):193-9. doi: 10.1159/000028794. PMID 10420129
- [Background] Graham T, Adams-Huet B, Gilbert N, Witthoff K, Gregory T, Walsh M. Effects of Initial Age and Severity on Cranial Remolding Orthotic Treatment for Infants with Deformational Plagiocephaly. J Clin Med. 2019 Jul 24;8(8):1097. doi: 10.3390/jcm8081097. PMID 31344968
- [Background] Pollack IF, Losken HW, Fasick P. Diagnosis and management of posterior plagiocephaly. Pediatrics. 1997 Feb;99(2):180-5. doi: 10.1542/peds.99.2.180. PMID 9024443
- [Background] Mottolese C, Szathmari A, Ricci AC, Ginguene C, Simon E, Paulus C. [Positional plagiocephaly: the place of cranial orthotics]. Neurochirurgie. 2006 Jun;52(2-3 Pt 2):184-94. doi: 10.1016/s0028-3770(06)71214-0. No abstract available. French. PMID 16981652
- [Background] Kim HY, Chung YK, Kim YO. Effectiveness of Helmet Cranial Remodeling in Older Infants with Positional Plagiocephaly. Arch Craniofac Surg. 2014 Aug;15(2):47-52. doi: 10.7181/acfs.2014.15.2.47. Epub 2014 Aug 14. PMID 28913190
- [Background] Cabrera-Martos I, Valenza MC, Valenza-Demet G, Benitez-Feliponi A, Robles-Vizcaino C, Ruiz-Extremera A. Effects of manual therapy on treatment duration and motor development in infants with severe nonsynostotic plagiocephaly: a randomised controlled pilot study. Childs Nerv Syst. 2016 Nov;32(11):2211-2217. doi: 10.1007/s00381-016-3200-5. Epub 2016 Jul 27. PMID 27465676
- [Background] Vles JS, Colla C, Weber JW, Beuls E, Wilmink J, Kingma H. Helmet versus nonhelmet treatment in nonsynostotic positional posterior plagiocephaly. J Craniofac Surg. 2000 Nov;11(6):572-4. doi: 10.1097/00001665-200011060-00010. PMID 11314498
- [Background] van Wijk RM, van Vlimmeren LA, Groothuis-Oudshoorn CG, Van der Ploeg CP, Ijzerman MJ, Boere-Boonekamp MM. Helmet therapy in infants with positional skull deformation: randomised controlled trial. BMJ. 2014 May 1;348:g2741. doi: 10.1136/bmj.g2741. PMID 24784879
- [Background] Kluba S, Kraut W, Calgeer B, Reinert S, Krimmel M. Treatment of positional plagiocephaly--helmet or no helmet? J Craniomaxillofac Surg. 2014 Jul;42(5):683-8. doi: 10.1016/j.jcms.2013.09.015. Epub 2013 Oct 15. PMID 24238984
- [Background] Kim SY, Park MS, Yang JI, Yim SY. Comparison of helmet therapy and counter positioning for deformational plagiocephaly. Ann Rehabil Med. 2013 Dec;37(6):785-95. doi: 10.5535/arm.2013.37.6.785. Epub 2013 Dec 23. PMID 24466513
- [Background] Wen J, Qian J, Zhang L, Ji C, Guo X, Chi X, Tong M. Effect of helmet therapy in the treatment of positional head deformity. J Paediatr Child Health. 2020 May;56(5):735-741. doi: 10.1111/jpc.14717. Epub 2019 Dec 23. PMID 31868272
- [Background] Lipira AB, Gordon S, Darvann TA, Hermann NV, Van Pelt AE, Naidoo SD, Govier D, Kane AA. Helmet versus active repositioning for plagiocephaly: a three-dimensional analysis. Pediatrics. 2010 Oct;126(4):e936-45. doi: 10.1542/peds.2009-1249. Epub 2010 Sep 13. PMID 20837585
- [Background] Clarren SK, Smith DW, Hanson JW. Helmet treatment for plagiocephaly and congenital muscular torticollis. J Pediatr. 1979 Jan;94(1):43-6. doi: 10.1016/s0022-3476(79)80347-9. PMID 758420
- [Background] Lam S, Pan IW, Strickland BA, Hadley C, Daniels B, Brookshier J, Luerssen TG. Factors influencing outcomes of the treatment of positional plagiocephaly in infants: a 7-year experience. J Neurosurg Pediatr. 2017 Mar;19(3):273-281. doi: 10.3171/2016.9.PEDS16275. Epub 2017 Jan 13. PMID 28084921
- [Background] Picart T, Beuriat PA, Szathmari A, Di Rocco F, Mottolese C. Positional cranial deformation in children: A plea for the efficacy of the cranial helmet in children. Neurochirurgie. 2020 Apr;66(2):102-109. doi: 10.1016/j.neuchi.2019.10.011. Epub 2020 Jan 17. PMID 31958410
- [Background] Lee HS, Kim SJ, Kwon JY. Parents' Perspectives and Clinical Effectiveness of Cranial-Molding Orthoses in Infants With Plagiocephaly. Ann Rehabil Med. 2018 Oct;42(5):737-747. doi: 10.5535/arm.2018.42.5.737. Epub 2018 Oct 31. PMID 30404423
- [Background] Demers L, Weiss-Lambrou R, Ska B. Development of the Quebec User Evaluation of Satisfaction with assistive Technology (QUEST). Assist Technol. 1996;8(1):3-13. doi: 10.1080/10400435.1996.10132268. PMID 10159726